CLINICAL TRIAL: NCT01588106
Title: Evaluation of the Impact of the CONTOUR® USB Blood Glucose Monitoring System With Integrated Data Management on Glycaemic Control in Insulin-treated Diabetic Patients
Brief Title: Evaluation of CONTOUR® USB BGMS on Glycaemic Control in Insulin-treated Diabetic Patients
Acronym: CONGO
Status: Completed | Type: Observational
Sponsor: GWT-TUD GmbH (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: GWT-2011-1
Record Dates: First submitted 2012-04-26; First posted 2012-04-30 (Estimated); Results first posted 2017-03-09 (Actual); Last update posted 2017-03-09 (Actual); Status verified 2016-01

CONDITIONS: Diabetes Mellitus Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Test group: patients using CONTOUR Next USB
- Control group: patients using standard CONTOUR

SUMMARY:
The purpose of this study is to evaluate if the use of the CONTOUR Next USB BGMS system with AutoLog and Trends features and integrated data management software (Glucofacts ™ DELUXE) enables behavioral changes that may lead to improvement in glycemic control, expressed as a reduction in HbA1c as primary endpoint.

Patients will be randomized either to using CONTOUR Next USB or CONTOUR. Patients will be trained in using the devices and return every 3 months until month 9 after baseline.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* Therapy with insulin only (ICT) or ICT in combination with Metformin
* HbA1c at baseline > 7.5% and < 11%
* Patients at least 18 years of age
* Patients willing to complete all study visits and study procedures including:

  * Testing their BG at least 3 times a day during the entire study.
  * Using the paper logbook provided (control group)
  * Using the Auto log meal-marker + reminder feature in CONTOUR Next USB regularly (TEST subjects only)
  * Using the Trends feature in CONTOUR Next USB regularly (TEST subjects only)
  * Uploading the CONTOUR Next USB meter to personal computer (subject must have personal computer at home or access to a computer - see system requirements in appendix for technical details).
* Patients who are able to speak, read and understand German
* Patients who are currently performing self-testing of blood glucose at home routinely (at least 3 times per day) for 4 weeks or more
* Patients who are currently adjusting there insulin dosages themselves based on the self-testing of blood glucose at home
* Written informed consent at beginning of the study

Exclusion Criteria:

* Patients who have been using CONTOUR Next USB meter regularly during the previous 12 months
* Patients treated with oral antidiabetic drugs except for Metformin; or diet alone
* Change of diabetes therapy within the last 3 months
* Change of HbA1c level of more than ±0.5% within the last 3 months
* Patients who are using a continuous blood glucose measurement system regularly
* Patients with home health aides who assist with their BG testing and /or insulin adjustment
* Patients with macroalbuminuria
* Steroid therapy within the last 3 months. Topic or inhalative use is no exclusion criterion when not used regularly (more than 5 times a week).
* Uncontrolled blood pressure ≥ 170/100 at screening
* BMI > 40 kg/m²
* Anemia according to WHO-definition (hemoglobin < 13 g/100 ml [male] or < 12 g/100 ml [female])
* Creatinin > 150 µmol/l and/or GFR < 50 mmol/min/ 1.73m² (measured within the last 3 months before screening)
* Operation with inpatient stay planned during the study
* Current pregnancy or pregnancy planned during the study; or breastfeeding women.
* Women with childbearing potential who are not practicing an acceptable method of birth control. Acceptable methods of birth control include tubal ligation, transdermal patch, intra uterine devices/systems (IUDs/IUSs), oral, implantable or injectable contraceptives, sexual abstinence, double barrier method and vasectomized partner
* Alcohol or drug abuse within the last 3 months
* Patients with the following impairments which, in the opinion of the investigator, would seriously compromise the integrity of the study:

  * Significant visual impairment
  * Significant hearing impairment
  * Cognitive disorder
  * Significant unstable co-morbidity (with notable change within the past 3 months)
  * Severe renal disease, disease with a strong impact on life expectancy
  * Inability to have or use and computer
  * Inability to use a meter correctly
  * Any other condition as per investigator's discretion
* Current participation in another clinical study. Participation in another trial within 6 weeks before screening.
* Employees of Bayer Vital Diabetes Care, the GWT or the University of Dresden

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients of assorted practices
Sampling Method: Probability Sample
Enrollment: 154 (Actual)
Dates: Start 2012-06; Primary Completion 2015-10 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Schwarz, Prof, Principal Investigator — Universitätsklinikum Carl Gustav Carus
Locations (16):
- Germany (16):
  - Diabetespraxis Prenzlauer Allee, Berlin
  - Praxis Dr. Fießelmann, Berlin
  - Praxis Dr. Stephan, Berlin
  - Gemeinschaftspraxis Lorra/Bonnermann, Bochum
  - Praxis Dr. Holderied, Brand-Erbisdorf
  - Spreewaldklinik, Burg
  - Diabeteszentrum DO, Dortmund
  - Studienzentrum Prof. Hanefeld, Dresden
  - Universitätsklinikum Dresden, Medizinische Klinik III, Dresden
  - Gemeinschaftspraxis Schaden, Düsseldorf
  - Praxis Dr. Stier, Freital
  - SMO.MD GmbH, Magdeburg
  - Praxis Dr. Ruhland, München
  - Metabolicum, München
  - Praxis Dr. Engelmayer, München
  - Diabeteszentrum Oschatz, Oschatz

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were screened and enrolled in 16 sites across Germany. Study start date was in June 2012 and recruitment was stopped in November 2014.
Groups:
- Test Group- CONTOUR Next USB: Subjects applied the CONTOUR NextT USB device. This group was not required to keep a paper log book. Subjects' blood glucose values were communicated to their health care professionals by using the data management software. Patients were trained in using the device and return every 3 months until month 9 after baseline.
- Control Group- Standard CONTOUR: Subjects used the standard CONTOUR device. Subjects' blood glucose values were communicated to their health care professionals via handwritten glucose log books. Patients were trained in using the device and return every 3 months until month 9 after baseline.
Period: Overall Study
Arm/Group | Test Group- CONTOUR Next USB | Control Group- Standard CONTOUR
Started | 78 | 76
Completed | 73 | 72
Not Completed | 5 | 4
Not completed — Withdrawal by Subject | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Test Group- CONTOUR Next USB | Control Group- Standard CONTOUR | Total
Number analyzed (Participants) | 73 | 72 | 145
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.10 (10.28) | 65.66 (9.08) | 63.87 (9.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 36 | 66
  Male | 43 | 36 | 79
HbA1c value at baseline [Mean (Standard Deviation); unit: %] | 8.61 (0.95) | 8.47 (0.97) | 8.54 (0.96)

OUTCOME MEASURES:

1. Primary Outcome: Reduction in HbA1c
Time Frame: Baseline, after 9 months
Population: All participants from whom HbA1c measurements were recorded at baseline and after 9 months.
Measure: Mean (Standard Deviation); unit: % (unit of HbA1c)
Arm/Group | Test Group- CONTOUR Next USB | Control Group- Standard CONTOUR
Number analyzed (Participants) | 58 | 56
% (unit of HbA1c) | -0.52 (0.83) | -0.14 (0.94)

ADVERSE EVENTS:
Arm/Group | Test Group- CONTOUR Next USB | Control Group- Standard CONTOUR
Serious Adverse Events (participants affected / at risk) | 0/78 | 1/76
Other Adverse Events (participants affected / at risk) | 13/78 | 9/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Test Group- CONTOUR Next USB (N=78) | Control Group- Standard CONTOUR (N=76)
severe thrombosis of the portal vein (Vascular disorders) | 0 (0) | 1 (1) — The patient suffered from severe thrombosis of the portal vein after Visit 1. This event was assessed as not being related to the trial Intervention but rather to the underlying concomitant disease(s).Patient was hospitalized but died in the end.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Test Group- CONTOUR Next USB (N=78) | Control Group- Standard CONTOUR (N=76)
Hypoglycaemia (Metabolism and nutrition disorders) | 13 (83) | 9 (106)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Publications or lectures on the findings of the present clinical trial either as a whole or at individual investigation sites must be approved by the sponsor in advance, and the sponsor reserves the right to review and comment on such documentation before publication.